CLINICAL TRIAL: NCT00150384
Title: Clinical Utility Of Caduet In Simultaneously Achieving Blood Pressure And Lipid Endpoints In A Specific Patient Population (CAPABLE)
Brief Title: Clinical Utility of Caduet in Achieving Blood Pressure and Lipid Endpoints in a Specific Patient Population
Acronym: CAPABLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3841025
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Hypertension; Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — amlodipine, atorvastatin drug combination

INTERVENTIONS:
Drug: Amlodipine/Atorvastatin

SUMMARY:
The purpose is to demonstrate the utility of Caduet (amlodipine/atorvastatin) in the African American population

ELIGIBILITY:
Inclusion Criteria:

* African American men and women with concurrent hypertension and dyslipidemia that is either treated or untreated
* Subjects must satisfy the blood pressure and LDL-C inclusion criteria for their respective Cardiovascular Risk group determined at screening

Exclusion Criteria:

* Subjects currently being treated with concomitant amlodipine and atorvastatin therapy, including Caduet
* Subjects with blood pressure at goal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-07; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of Caduet therapy by assessing the percentage of intent-to-treat subjects achieving both BP and lipid treatment goals (JNC VII and NCEP ATP III)

SECONDARY OUTCOMES:
To assess the percentage of subjects achieving treatment goals(JNC VII and NCEP) stratified by the final BP and lipid therapy doses, respectively, the change from baseline in lipid profile, SBP and DBP

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (76):
- United States (76):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Oakland, California
  - Pfizer Investigational Site, Pico Rivera, California
  - Pfizer Investigational Site, Bridgeport, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Aventura, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Vero Beach, Florida
  - Pfizer Investigational Site, Athens, Georgia
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Columbus, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Lincolnton, Georgia
  - Pfizer Investigational Site, Savannah, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Maywood, Illinois
  - Pfizer Investigational Site, Merrillville, Indiana
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Bossier City, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Columbia, Maryland
  - Pfizer Investigational Site, Randallstown, Maryland
  - Pfizer Investigational Site, Rockville, Maryland
  - Pfizer Investigational Site, Westminster, Maryland
  - Pfizer Investigational Site, Brockton, Massachusetts
  - Pfizer Investigational Site, Wellesley Hills, Massachusetts
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Lansing, Michigan
  - Pfizer Investigational Site, Livonia, Michigan
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Cherry Hill, New Jersey
  - Pfizer Investigational Site, East Orange, New Jersey
  - Pfizer Investigational Site, Elizabeth, New Jersey
  - Pfizer Investigational Site, Hammonton, New Jersey
  - Pfizer Investigational Site, South Bound Brook, New Jersey
  - Pfizer Investigational Site, Voorhees Township, New Jersey
  - Pfizer Investigational Site, Woodbury, New Jersey
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Mineola, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Greenville, North Carolina
  - Pfizer Investigational Site, Monroe, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Maumee, Ohio
  - Pfizer Investigational Site, Perrysburg, Ohio
  - Pfizer Investigational Site, Bensalem, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Bamberg, South Carolina
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Clinton, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Simpsonville, South Carolina
  - Pfizer Investigational Site, Bartlett, Tennessee
  - Pfizer Investigational Site, Jackson, Tennessee
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Emporia, Virginia
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Milwaukee, Wisconsin